CLINICAL TRIAL: NCT07006350
Title: Heart Failure and Therapeutic Education
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Gonesse (Other)
Responsible Party: Sponsor
Other Study IDs: 0105_URC
Record Dates: First submitted 2025-05-28; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Heart Failure; Health Education; Diet, Sodium-Restricted; Disease Management; Therapeutics
MeSH Terms: conditions — Heart Failure; Health Education

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study looks at whether a special program called the Heart Failure Therapeutic Education Unit (UTIC) helps reduce hospital stays for people with heart failure. It is a retrospective study, which means we are looking back at the records of patients who were followed at the UTIC in 2023 and 2024.

We want to find out two things:

If patients who followed the UTIC program were hospitalized less often.

If the advice they received-especially about diet-helped improve their condition.

Only adult patients who were treated at the UTIC are included in the study. We will not use data from patients who are under 18, were not treated in UTIC, or did not give permission to use their information.

The study takes place over two weeks, from March 24 to April 6, 2025.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age ≥ 18 years)
* Patients diagnosed with heart failure
* Patients followed in the Heart Failure Therapeutic Education Unit (UTIC) at the General Hospital (CHG)
* Follow-up occurred during the years 2023 or 2024

Exclusion Criteria:

* Patients who do not consent to the use of their medical data
* Minors (under 18 years old)
* Patients not followed in the UTIC program

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants will be selected from adult patients diagnosed with heart failure who received care at the Heart Failure Therapeutic Education Unit (UTIC) of the General Hospital (CHG). The population includes patients who were followed by the UTIC during the years 2023 and 2024. Only those who meet the inclusion criteria and do not fall under the exclusion criteria (e.g., minors, non-UTIC patients, or those who oppose the use of their data) will be considered for the study.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2025-03-24 (Actual); Primary Completion 2025-04-06 (Actual); Study Completion 2025-04-06 (Actual)

PRIMARY OUTCOMES:
Number of hospitalizations among patients with heart failure who were followed at the Unité Thérapeutique de l'Insuffisance Cardiaque (UTIC). | Review of hospital records for patients seen in 2023-2024.

CONTACTS AND LOCATIONS:
Locations (1):
- France, Gonesse, France, France